CLINICAL TRIAL: NCT06563570
Title: The Effect of Teleyoga on Balance, Frailty, Cognition and Quality of Life in Liver Transplant Patients
Brief Title: The Effect of Teleyoga in Liver Transplant Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Bilge Summakoğlu, physiotherapist, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEU-SBF-BS-01
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplant Disorder
Keywords: liver transplantation; yoga; balance; cognition
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Other): The only group in the study was liver transplant patients who practised yoga online.
  Interventions: Other: yoga (online)

INTERVENTIONS:
Other: yoga (online) — 8-week online yoga practices, 2 days a week

SUMMARY:
Online yoga practices will be applied in liver transplant patients and the effects of online yoga on balance, frailty, cognition and quality of life of transplant patients will be examined.

DETAILED DESCRIPTION:
The study will include liver transplant patients who applied to Dokuz Eylül University Faculty of Medicine, Department of Surgical Medical Sciences, Department of General Surgery Outpatient Clinic. The aim of the study is to investigate the effect of online yoga practice on balance, frailty, cognition and quality of life levels in liver transplant patients. The study will include 26 patients with liver transplantation who meet the criteria. Participants will first be informed about the study and individuals will be included in the study after signing the informed consent form. Demographic information of liver transplant patients will be obtained and their balance, frailty, cognition and quality of life levels and post-transplant symptoms (symptoms seen in people) will be evaluated.

Online yoga practices will be applied to liver transplant patients for 8 weeks, 2 days a week, 30 minutes a day. Online yoga (teleyoga) will be performed via video call with people who meet the inclusion criteria. After 8 weeks of yoga intervention, balance, frailty, cognition and quality of life levels and post-transplant symptoms will be re-evaluated.

Balance measurements will be evaluated with Biodex Balance System (BSS). Frailty levels will be assessed by Short Physical Performance Battery and FRAIL frailty questionnaire. Cognition will be assessed by trail making test and stroop test. Quality of life will be evaluated with Short Form-36 quality of life scale and post-transplantation symptoms will be evaluated with Modified Post-Transplantation Symptom Occurrence and Discomfort Status-58-Item Scale-Turkey.

The evaluations are planned to last 1-2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Liver transplantation at least 6 months ago
* Individuals with a Mini Mental Test score greater than 24

Exclusion Criteria:

* Pregnancy
* Central Nervous System Dysfunction
* Musculoskeletal deformity
* Vestibular dysfunction
* Specific neurological pathology (Parkinson's, stroke, epilepsy)
* Those with severe systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-09-16 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System | two weeks
  Balance will be assessed separately with the Biodex Balance System (Biodex Medical Systems, Inc., Shirley, NY) standing, eyes open, static and dynamic. For static and dynamic balance assessments, each test will be performed for 20 seconds with 3 repetitions. Average scores will be recorded after the evaluation. An increase in scores indicates worsening of balance and a decrease in scores indicates improvement in balance.

SECONDARY OUTCOMES:
FRAIL frailty scale | two weeks
  In the FRAIL frailty scale; patients' weight loss, fatigue, slowness, decreased physical activity and weakness are examined. Those with 0 points from this questionnaire are classified as fit, those with 1-2 points are classified as pre-frail, and those with 3 or more points are classified as frail.
Short Physical Performance Battery | two weeks
  And The Short Physical Performance Battery consists of 3 objective tests assessing lower body function. All three physical performance measures (walking speed, balance, getting up from a chair) are scored between 0-4 according to the duration of the activity, and the scores of the three tests are summed to obtain a total score between 0 ( bad) and 12 (very good).
The stroop test | two weeks
  The Stroop test . On each card, there are 6 lines consisting of 4 items. These stimulus cards constitute the parts of the test and the tasks that the participant has to fulfil against these stimulus cards constitute the parts of the test.
the tracking test | two weeks
  There are two parts in the test, A and B. The completion time of the sequential patterns in the sections is analysed. Eight sub-scores are calculated by looking at the time, number of errors and corrections.
Modified Transplantation Symptom Occurrence and Discomfort - 58-Item Scale | two weeks
  Each item of the scale assesses a side effect of immunosuppressive drugs. The form assesses the frequency or intensity of symptom occurrence and the discomfort caused by the symptom in the presence of the symptom. People will be asked to tick '0' if they have not experienced any symptoms in the last 4 weeks, '1' if they have rarely, '2' if they have sometimes, '3' if they usually, or '4' if they have experienced a lot of symptoms. Afterwards, according to the distress caused by the symptom, the respondent will be asked to mark the situation he/she experienced from 0 (no distress at all) to 4 (extreme distress).
short form-36 quality of life scale | two weeks
  It was evaluated with Short form-36 quality of life scale. It evaluates quality of life especially in individuals with physical illness and provides measurement of quality of life in 8 dimensions: physical function (10 items), social function (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), vitality (4 items), pain (2 items) and general perception of health (5 items). A total score is given separately for each subscale and scores range from 0-100. A score of '100' indicates good health status, while a score of '0' indicates poor health status.
Beck depression scale | two weeks
  Depression assessment with Beck depression scale. The scale consists of 21 items. Each item is scored between 0-3. A higher total score indicates a higher severity or level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: bilge summakoğlu, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)